CLINICAL TRIAL: NCT03329755
Title: Optimization of the Patient Care Pathway in Immuno-oncology
Acronym: OPTIMMUNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16 CUTA 05
Record Dates: First submitted 2017-10-25; First posted 2017-11-06 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Melanoma
Keywords: Advanced melanoma; Immune checkpoint; E-follow-up
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Other: Dedicated and coordinated e-follow-up during the treatment period
- Standard (Other)
  Interventions: Other: Standard follow-up during the treatment period

INTERVENTIONS:
Other: Dedicated and coordinated e-follow-up during the treatment period — * Completion of questionnaires using an electronic tool
  * Telephone follow-up between the nurse and the patient
  * Completion of the Quality of Life Questionnaire Core 30 (QLQ-C30)
  Arms: Experimental
Other: Standard follow-up during the treatment period — - Completion of the Quality of Life Questionnaire Core 30 (QLQ-C30)
  Arms: Standard

SUMMARY:
This study compares the care pathway of melanoma patients treated by immunotherapy in two ambulatory care structures. The aim is to measure if a care structure specialized in immuno-oncology could rationalize the care of patients.

This protocol will be based on two different follow-up during the treatment period:

* dedicated and coordinated e-follow-up (IUCT-O in Toulouse)
* standard follow-up (University Hospital Center in Bordeaux)

Patients will be followed from the first cycle of immunotherapy until 3 months after the initiation treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with advanced (unresectable melanoma (stage III)) or metastatic (stage IV) melanoma and starting an Immune Checkpoint Inhibitor treatment (Monotherapy or Combination Therapy)
2. Patient starting first cycle of Immune Checkpoint Inhibitor treatment in an ambulatory care structure
3. Treatment which can be delayed for 7 days or more
4. Age > or = 18 years old
5. Patient with a phone and/or computer equipment
6. Patient affiliated to the french social security system
7. Patient must provide written informed consent prior to any study-specific procedure or assessment

Exclusion Criteria:

1. Patient with diagnosis other than advanced melanoma
2. Patient who must receive a treatment other than Immune Checkpoint Inhibitor
3. Treatment administered during a conventional hospital stay (period of more than 24 hours)
4. Patient with no caregiver
5. Pregnant or breastfeeding women
6. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
7. Patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Average length of administrative stay in the hospital | 3 months by patient

SECONDARY OUTCOMES:
Number of cancelled or delayed hospital stay | 3 months by patient
Patient quality of life using the Quality of Life Questionnaire Core 30 (QLQ-C30) | 3 months by patient
Treatment response rate at 3 months | 3 months by patient
Correlation between the day hospital stay and the patient general health | 3 months by patient
Frequency of web interface completion (Experimental arm only) | 3 months by patient
Patient satisfaction to the e-follow-up (Experimental arm only) | 3 months by patient
Rate of reclassified alerts after intervention of nurse (Experimental arm only) | 3 months by patient

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Saint André, CHU de Bordeaux, Bordeaux
  - Institut claudius regaud IUCT ONCOPOLE, Toulouse